CLINICAL TRIAL: NCT00949962
Title: Immediate or Early Salvage Post-operative External Radiotherapy Combined With Concomitant and Adjuvant Hormonal Treatment Versus Immediate or Early Salvage Postoperative External Radiotherapy Alone in pT3a-b R0-1 cN0M0 / pT2R1 cN0M0, Gleason Score 5-10 Prostatic Carcinoma. A Phase III Study
Brief Title: Post-operative or Early Salvage XRT and ADT for High Risk PCa
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poorly recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-22043-30041; EU-20950; 2006-002772-17 (EudraCT Number)
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Leuprolide; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients undergo post-operative conformal external beam irradiation for 6.5 weeks.
  Interventions: Radiation: 3-dimensional conformal radiation therapy
- Arm II (Experimental): Beginning on day -5 to -3, patients receive an antiandrogen for 2-4 weeks. Beginning on day 0, patients receive leuprolide acetate subcutaneously once (6-month depot) and undergo conformal external beam irradiation 5 times weekly for 6.5 weeks.
  Interventions: Drug: antiandrogen therapy; Drug: leuprolide acetate; Radiation: 3-dimensional conformal radiation therapy

INTERVENTIONS:
Drug: antiandrogen therapy — Given systemically
  Arms: Arm II
Drug: leuprolide acetate — Given subcutaneously
  Arms: Arm II
Radiation: 3-dimensional conformal radiation therapy — Undergo radiotherapy

SUMMARY:
RATIONALE: Conformal radiation therapy uses a 3-dimensional (3-D) image of the tumor to help focus thin beams of radiation directly on the tumor. Giving conformal external-beam radiation therapy in higher doses over a shorter period of time may kill more tumor cells and have fewer side effects. Androgens can cause the growth of prostate cancer cells. Hormone therapy, such as leuprolide acetate, may lessen the amount of androgens made by the body. It is not yet known whether radiation therapy is more effective when given together with or without hormone therapy in treating patients with prostate cancer who have undergone surgery.

PURPOSE: This randomized phase III trial is studying radiation therapy to see how well it works compared with radiation therapy given together with hormone therapy in treating patients who have undergone surgery for stage I, stage II, or stage III prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate the potential benefit of post-operative radiotherapy with vs without a combined and adjuvant treatment consisting of short-term androgen suppression for improving the biochemical progression-free survival of patients who have undergone radical prostatectomy for stage I-III prostate cancer.

OUTLINE: This is a multicenter study. Patients are stratified according to institution, pathological stage (pT2R1 vs pT3R0 vs pT3R1), Gleason sum (≤ 3+4 vs ≥ 4+3), and WHO performance status (0 vs 1). Within 3 months after radical surgery, patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo post-operative conformal external beam irradiation for 6.5 weeks.
* Arm II: Beginning between days -5 to -3, patients receive an antiandrogen for 2-4 weeks. Beginning on day 0, patients receive leuprolide acetate subcutaneously once (6-month depot) and undergo conformal external beam irradiation 5 times weekly for 6.5 weeks.

Patients undergo quality of life assessments periodically.

After completion of study treatment, patients are followed up every 6 months for 5 years and then yearly thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of prostate cancer

  * Clinical stage cT1-2-3a, N0, M0 disease pre-operatively
  * Pre-operative PSA ≤ 5 x upper limit of normal
* Presenting the following conditions after radical prostatectomy:

  * Gleason sum 5-10
  * Pathologic stage pT2R1 (positive surgical margins with at least a tumor trans-section > 2 mm) or pT3a-b (irrespective of margin status)
  * Negative lymph node (LN) status (pN0) by LN sampling or LN dissection

    * Unknown pathological LN status is not allowed, except for disease classified as cT ≤ cT1c with baseline PSA ≤ 10 ng/mL, Gleason score < 7, and ≥ 12 positive core biopsies < 50%
  * Undetectable post-operative PSA within 3 months of surgery

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* WBC ≥ 3 x 10^9/L
* Hemoglobin ≥ 110 g/L
* Platelet count ≥ 100 x 10^9/L
* No other malignancy except adequately treated basal cell carcinoma of the skin or other malignancy from which the patient has been disease free for at least 5 years
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 5 years since prior chemotherapy
* No prior pelvic irradiation
* No prior bilateral orchiectomy
* No prior hormonal treatment except neoadjuvant treatment lasting ≤ 3 months
* No other concurrent anticancer agent or modality

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Biochemical progression-free survival

SECONDARY OUTCOMES:
Clinical progression-free survival
Distant-metastases-free survival
Overall survival
Quality of life as assessed by QLQ-C30 and QLQ-PR25 at baseline and at 6 months, 1 year, 2 years, and 5 years after treatment
Acute and late toxicity according to NCI CTCAE version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bolla, MD, Principal Investigator — CHU de Grenoble - Hopital de la Tronche
Locations (1):
- European Organization for Research and Treatment of Cancer, Grenoble, France